CLINICAL TRIAL: NCT01500837
Title: Treatment of Methicillin-sensitive Staphylococcus Aureus Orthopaedic Infections With Clindamycin in Combination With Rifampin or Levofloxacin: a Randomized Pharmacological and Clinical Study (the CLINDOS Trial)
Brief Title: Treatment of Methicillin-sensitive Staphylococcus Aureus (MSSA)
Acronym: CLINDOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K000000
Record Dates: First submitted 2011-11-28; First posted 2011-12-29 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2010-09

CONDITIONS: Osteoarticular Infection
Keywords: Staphylococcus aureus; osteoarticular infection; clindamycin; serum concentration; orthopedic surgery
MeSH Terms: conditions — Staphylococcal Infections | interventions — Clindamycin; Rifampin; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIFAMPIN (Active Comparator): CLINDAMYCIN + RIFAMPIN
  Interventions: Drug: association of RIFAMPIN + CLINDAMYCIN
- LEVOFLOXACIN (Active Comparator): CLINDAMYCIN + LEVOFLOXACIN
  Interventions: Drug: association of LEVOFLOXACIN+ CLINDAMYCIN

INTERVENTIONS:
Drug: association of RIFAMPIN + CLINDAMYCIN — association of RIFAMPIN + CLINDAMYCIN
  Other Names: RIFAMPIN
  Arms: RIFAMPIN
Drug: association of LEVOFLOXACIN+ CLINDAMYCIN — association of LEVOFLOXACIN+ CLINDAMYCIN
  Other Names: LEVOFLOXACIN
  Arms: LEVOFLOXACIN

SUMMARY:
Background:

One of the leading causes of peri-operative osteoarticular infections (OAI) is Staphylococcus aureus. Treatment usually requires surgical debridement in association with appropriate antibiotic therapy. After surgery, an intravenous (IV) antibiotic therapy is routinely indicated for 10 to 15 days, followed by a minimal one-month oral treatment. In this protocol, the latter includes clindamycin in combination with rifampin or levofloxacin. Clindamycin is considered a good option in staphylococcal infections, because of its action against biofilm formation and bacterial adherence, its high level of joint and bone penetration and its good tolerance. Rifampin, a potent cytochrome P-450 inducer, enhances the elimination of a large number of drugs. Therefore, an influence of rifampin on clindamycin pharmacokinetics must be considered.

Objectives:

The primary objective is to compare the influence of rifampin and levofloxacin respectively on the pharmacokinetics of clindamycin in a randomized series of peri-operative staphylococcal OAI. The investigators then seek to determine the optimal drug association with regard to infection control and drug tolerance.

Study design:

Monocentric, randomized, open label, comparative study

Study period:

From November 2010 to October 2011.

Materials and Methods:

Following surgical debridement and after 10 to 15 days of IV antibiotherapy, patients are randomly assigned either to the "clindamycin/rifampin" arm either to the "clindamycin/levofloxacin" arm, according to the antimicrobial susceptibility testing. Peak and trough serum concentrations of clindamycin are measured at day-1, day-15 and day-30 of oral treatment. Rifampin and levofloxacin serum concentrations are measured at the same intervals to monitor patient compliance.

DETAILED DESCRIPTION:
Background:

One of the leading causes of peri-operative osteoarticular infections (OAI) is Staphylococcus aureus. Treatment usually requires surgical debridement in association with appropriate antibiotic therapy. After surgery, an intravenous (IV) antibiotic therapy is routinely indicated for 10 to 15 days, followed by a minimal one-month oral treatment. In this protocol, the latter includes clindamycin in combination with rifampin or levofloxacin. Clindamycin is considered a good option in staphylococcal infections, because of its action against biofilm formation and bacterial adherence, its high level of joint and bone penetration and its good tolerance. Rifampin, a potent cytochrome P-450 inducer, enhances the elimination of a large number of drugs. Therefore, an influence of rifampin on clindamycin pharmacokinetics must be considered.

Objectives:

The primary objective is to compare the influence of rifampin and levofloxacin respectively on the pharmacokinetics of clindamycin in a randomized series of peri-operative staphylococcal OAI. The investigators then seek to determine the optimal drug association with regard to infection control and drug tolerance. Study design: monocentric, randomized, open label, comparative study

Study period:

From November 2010 to October 2011.

Materials and Methods:

Following surgical debridement and after 10 to 15 days of IV antibiotherapy, patients are randomly assigned either to the "clindamycin/rifampin" arm either to the "clindamycin/levofloxacin" arm, according to the antimicrobial susceptibility testing. Peak and trough serum concentrations of clindamycin are measured at day-1, day-15 and day-30 of oral treatment. Rifampin and levofloxacin serum concentrations are measured at the same intervals to monitor patient compliance. Infection cure is evaluated clinically, with periodic X-rays and CRP dosage in serum.

ELIGIBILITY:
Inclusion Criteria:

* subject over 18 years with a IOA with GERME sensitivity to three antibiotics,
* Patient in orthopedic unit of HEGP,
* Patient who received and understood the information and who signed consent,

Exclusion Criteria:

* Known allergy to one of three antibiotics and / or excipients,
* Pregnancy or during lactation,
* Congenital galactosemia, malabsorption of glucose and galactose, or lactase deficiency,
* History of tendinopathy with fluoroquinolones,
* G6PD deficiency,
* porphyria,
* subject receiving a protease inhibitor,
* subject receiving anticoagulants
* Malabsorption syndrome,
* subject unable to follow the protocol (organizational problem, intellectual disability, ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Measurement of peak and trough serum concentrations of clindamycin | 1 month
  Measurement of peak and trough serum concentrations of clindamycin will be performed at Day 1, Day 15 and Day 30

SECONDARY OUTCOMES:
proportion of patients healing (as determined from absence of fever, absence of pain and favorable aspect of scar). | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Sabatier, PD, PhD, Study Director — Department of Pharmacology
Locations (1):
- Assistance Publique Hopitaux de Paris, Paris, France

REFERENCES:
- [Derived] Bernard A, Kermarrec G, Parize P, Caruba T, Bouvet A, Mainardi JL, Sabatier B, Nich C. Dramatic reduction of clindamycin serum concentration in staphylococcal osteoarticular infection patients treated with the oral clindamycin-rifampicin combination. J Infect. 2015 Aug;71(2):200-6. doi: 10.1016/j.jinf.2015.03.013. Epub 2015 Apr 30. PMID 25936632